CLINICAL TRIAL: NCT03158883
Title: UCDCC#270: A Pilot Study of Avelumab and Stereotactic Ablative Radiotherapy in Non-responding and Progressing NSCLC Patients Previously Treated With a PD-1 Inhibitor
Brief Title: UCDCC#270: Avelumab and Stereotactic Ablative Radiotherapy in Non-responding and Progressing NSCLC Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Megan Daly, MD (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor-Investigator, Megan Daly, MD, Assistant Professor, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1054028; UCDCC#270 (Other: UC Davis IRB)
Record Dates: First submitted 2017-05-08; First posted 2017-05-18 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Non-small Cell Lung Cancer (NSCLC)
Keywords: Avelumab; NSCLC; Stereotactic ablative radiotherapy (SAR)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — avelumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Two groups (n=13) of non-responders and progressors will go through the same treatment regime.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Non-responders (Experimental): Patients who initially progress at first response assessment on a PD-1 inhibitor will be enrolled to the "non-responder" arm.
  * Avelumab: 10 mg/kg administered by IV infusion q2w (1 cycle = 14 [±2] days).
  * Stereotactic ablative radiotherapy (SAR): the prescription dose will be 50 Gy over 5 fractions of 10 Gy each on an every 2 day basis (i.e., 2-3 treatments per week, with a minimum of 40 hours and a maximum of 96 hours between treatments) and completed within 1.5-2 weeks. SAR treatment will not be repeated.
  Interventions: Drug: Avelumab; Radiation: Stereotactic ablative radiotherapy (SAR)
- Progressors (Experimental): Patients who initially present with PR, CR, or SD to a PD-1 inhibitor but subsequently progress will be enrolled to the "progressor" arm.
  * Avelumab: 10 mg/kg administered by IV infusion q2w (1 cycle = 14 [±2] days).
  * Stereotactic ablative radiotherapy (SAR): the prescription dose will be 50 Gy over 5 fractions of 10 Gy each on an every 2 day basis (i.e., 2-3 treatments per week, with a minimum of 40 hours and a maximum of 96 hours between treatments) and completed within 1.5-2 weeks. SAR treatment will not be repeated.
  Interventions: Drug: Avelumab; Radiation: Stereotactic ablative radiotherapy (SAR)

INTERVENTIONS:
Drug: Avelumab — Avelumab: 10 mg/kg administered by IV infusion q2w (1 cycle = 14 [±2] days).
  Other Names: anti-PD-L1 IgG1 monoclonal antibody
Radiation: Stereotactic ablative radiotherapy (SAR) — SAR: the prescription dose will be 50 Gy over 5 fractions of 10 Gy each on an every 2 day basis (i.e., 2-3 treatments per week, with a minimum of 40 hours and a maximum of 96 hours between treatments) and completed within 1.5-2 weeks. SAR treatment will not be repeated.
  Other Names: stereotactic body radiotherapy; SBRT; SAR

SUMMARY:
This is a pilot, single center, open-label study to examine the ORR, safety, and toxicity of avelumab in combination with SAR in non-responding and progressing NSCLC patients previously treated with a PD-1 Inhibitor.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer deaths worldwide. More than half of lung cancer patients present with metastatic disease at diagnosis, with a median survival of only 10-12 months. In recent years the development of more efficacious therapies for metastatic non-small cell lung cancer (NSCLC) based upon an improved understanding of the underlying tumor biology has resulted in an improvement in median overall survival by several months. However, survival remains poor for most patients and there remains an urgent unmet need for novel treatment strategies to improve survival for these patients.

Avelumab is a fully human anti-PD-L1 IgG1 monoclonal antibody. In phase I studies, avelumab was well-tolerated at a dose of 10 mg/kg IV Q2 weeks with the most frequently observed treatment related adverse events including fatigue, infusion-related reactions, nausea, chills, diarrhea, and pyrexia. However, many patients will not respond to checkpoint inhibition, and developing strategies to further improve the efficacy and extend the benefit of these treatments to non-responding and progressing patients is an area of substantial need. Among NSCLC patients, approximately 80% of patients will not respond to a checkpoint inhibitor as monotherapy.

Combinatorial strategies may increase response rates. Radiotherapy is an intriguing partner therapy, with preclinical and clinical studies confirming the immunomodulatory effects of radiotherapy. There is particularly interest in the use of radiotherapy in patients who have failed a checkpoint inhibitor as monotherapy as this approach will isolate the effects of radiation in enhancing response rates.

Stereotactic ablative radiotherapy (SAR) (also known as stereotactic body radiotherapy or SBRT) has emerged as a potentially curative treatment option for patients with early stage, medically inoperable non-small cell lung cancer and as a safe and effective local treatment for metastatic lesions.

The investigators hypothesize that local radiotherapy can augment the systemic effects of avelumab in NSCLC patients previously refractory to a checkpoint inhibitor previously used as standard-of-care treatment. This proposal seeks to gain insight into the clinical and biological efficacy of this combination.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Ability to comply with the protocol.
3. Adults >18 years of age with histologically proven stage IV non-small cell lung cancer.
4. At least two sites of measurable disease as defined by RECIST 1.1; one of which must be amenable to treatment with SAR and accessible for a mandatory pre-treatment biopsy and a post- treatment biopsy at physician discretion. If a pulmonary nodule is being considered for SAR it must range in size from 1-5 cm.
5. Have provided written consent for protocol directed biopsies.
6. Patients with treated supratentorial metastases are allowed if stable, the patient is off steroids or on a stable or decreasing dose of ≤10 mg daily prednisone (or equivalent) and no evidence of intracranial hemorrhage.
7. Archival tumor sample available. A minimum of 10 unstained slides. No fine needle aspiration (FNAs) allowed or tumor tissue from bone.
8. ECOG performance status score of 0 or 1 (Appendix 1).
9. Life expectancy ≥ 3 months.
10. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days of the first study treatment:

    1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused)
    2. Liver function tests meeting the following criteria: total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 × ULN (for subjects with documented metastatic disease to the liver).
    3. INR and aPTT <1.5 × ULN (for patients on anticoagulation they must be receiving a stable dose for at least 1 week prior to randomization)
    4. Creatinine clearance >30 mL/min by Cockcroft-Gault formula (or local institutional standard method).
11. No history of severe hypersensitivity reactions to other mAbs.
12. No other active malignancy.
13. No active autoimmune disease or a history of known or suspected autoimmune disease except as detailed in the exclusion criteria below.
14. No chemotherapy or radiotherapy within the past 28 days.
15. Any number of prior treatments is allowed. Must have failed at least one treatment regimen for metastatic disease and must have failed platinum-based chemotherapy (including as treatment for localized disease) or be deemed ineligible for platinum-based therapy by the treating medical oncologist.
16. Most recent prior regimen was a PD-1 inhibitor (nivolumab or pembrolizumab) with progression. Last dose must have been delivered within 90 days of enrollment.
17. Highly effective contraception for both male and female subjects if the risk of conception exists. (Note: The effects of the trial drug on the developing human fetus are unknown; thus, women of childbearing potential and men able to father a child must agree to use 2 highly effective contraception, defined as methods with a failure rate of less than 1% per year. Highly effective contraception is required at least 28 days prior, throughout and for at least 60 days after avelumab treatment.
18. Negative serum pregnancy test at screening for women of childbearing potential.

Exclusion Criteria:

1. Patients whose tumors contain activating EGFR mutations or ALK rearrangement should be excluded from this study, unless disease has progressed on all available, approved therapies targeting the EGFR mutation or ALK rearrangement.
2. All subjects with brain metastases, except those meeting the following criteria:

   1. Brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to enrollment
   2. No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
   3. Subjects must be either off steroids or on a stable or decreasing dose of <10mg daily prednisone (or equivalent)
3. Leptomeningeal disease.
4. Uncontrolled pleural or pericardial effusion or ascites that would require recurrent drainage.
5. Uncontrolled tumor related pain.
6. Uncontrolled hypercalcemia.
7. Pregnant and lactating women.
8. Uncontrolled concomitant disease.
9. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
10. Significant acute or chronic infections including, among others:

    1. Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
    2. Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive)
11. Oral or IV antibiotics within 2 weeks prior to enrollment.
12. Active tuberculosis
13. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI CTCAE v 4.03), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma).
14. Known hypersensitivity or allergy to any component of the avelumab formulation.
15. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

    1. Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
    2. Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day
    3. Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable
16. Patients with a prior allogeneic bone marrow transplantation or prior solid organ transplantation.
17. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan. A history of radiation pneumonitis in the radiation field (fibrosis) is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 90 days after completion of study treatment
  Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 90 days after completion of study treatment.
  OS is defined as the duration of time from the start of treatment to death from any cause.
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 90 days after completion of study treatment.
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Disease Control Rate (DCR) | From date of randomization to end of study, assessed up to 90 days follow-up
  DCR is defined as the percentage of patients that achieve an objective tumor response or stable disease to therapy.
Duration of Stable Disease | From date of randomization to end of study, assessed up to 90 days follow-up
  SD is measured from the start of the treatment until the criteria for disease progression are met, taking as reference the smallest measurements recorded since the treatment started.
Duration of Overall Response | From date of randomization to end of study, assessed up to 90 days follow-up
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that recurrence or PD is objectively documented, taking as reference for PD the smallest measurements recorded since the treatment started.
Confirmation | From date of randomization to end of study, assessed up to 90 days follow-up
  The main goal of confirmation of objective response is to avoid overestimating the response rate observed. In cases where confirmation of response is not feasible, it should be made clear when reporting the outcome of such studies that the responses are not confirmed.
Immune Related Response Criteria | From date of randomization to end of study, assessed up to 90 days follow-up
  A growing body of literature indicates that radiographic responses to immunotherapy may have different patterns and kinetics than what would be expected with traditional cytotoxic therapies. To account for these differences we will also characterize radiographic outcomes using the immune related response criteria outlined by Wolchok and colleagues as an exploratory outcomes.
Evaluation of Best Overall Response | From date of randomization to end of study, assessed up to 90 days follow-up
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). In general, the patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Daly, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No